CLINICAL TRIAL: NCT01955837
Title: Randomized, Double-Blind, Phase III Study of TAS-102 Versus Placebo in Asian Patients With Metastatic Colorectal Cancer Refractory or Intolerable to Standard Chemotherapies
Brief Title: Study of Trifluridine/Tipiracil (TAS-102) in Patients With Metastatic Colorectal Cancer in Asia
Acronym: TERRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10040090
Record Dates: First submitted 2013-09-19; First posted 2013-10-08 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- TAS-102 (Experimental)
  Interventions: Drug: TAS-102
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAS-102 — TAS-102 (35 mg/m2/dose) orally, twice daily on days 1-5 and 8-12 of each 28-day cycle. Number of cycles: until at least one of the discontinuation criteria is met.
  Arms: TAS-102
Drug: Placebo — Placebo orally, twice daily on days 1-5 and 8-12 of each 28-day cycle. Number of cycles: until at least one of the discontinuation criteria is met.
  Arms: Placebo

SUMMARY:
To compare the effects of TAS-102 with placebo in patients with metastatic colorectal cancer refractory or intolerable to standard chemotherapies.

DETAILED DESCRIPTION:
This is a multinational, double-blind, two-arm, parallel, randomized Phase 3 comparison study evaluating the efficacy and safety of TAS-102 versus placebo in patients with refractory metastatic colorectal cancer. Patients will be randomly assigned (2:1) to TAS-102 (experimental arm) or placebo (control arm).

ELIGIBILITY:
Inclusion Criteria:

* Has provided written informed consent
* Has adenocarcinoma of the colon or rectum
* Has failed at least 2 prior regimens of standard chemotherapies for metastatic colorectal cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Is able to take medication orally
* Has adequate organ function (bone marrow, kidney and liver)
* Women of childbearing potential must have a negative pregnancy test and must agree to adequate birth control if conception is possible. Males must agree to adequate birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2013-09; Primary Completion 2016-02-16 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- China (2):
  - Peking University Cancer Hospital, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai
- Asan Medical Center, Seoul, South Korea
- Chulalongkorn University & The King Chulalongkorn Memorial Hospital, Bangkok, Thailand

REFERENCES:
- [Derived] Xu J, Kim TW, Shen L, Sriuranpong V, Pan H, Xu R, Guo W, Han SW, Liu T, Park YS, Shi C, Bai Y, Bi F, Ahn JB, Qin S, Li Q, Wu C, Ma D, Lin D, Li J. Results of a Randomized, Double-Blind, Placebo-Controlled, Phase III Trial of Trifluridine/Tipiracil (TAS-102) Monotherapy in Asian Patients With Previously Treated Metastatic Colorectal Cancer: The TERRA Study. J Clin Oncol. 2018 Feb 1;36(4):350-358. doi: 10.1200/JCO.2017.74.3245. Epub 2017 Dec 7. PMID 29215955

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 406 centers in China, the Republic of Korea and Thailand from 16 October 2013 to 15 June 2015.
Groups:
- TAS-102（Trifluridine/Tipiracil）: Trifluridine/Tipiracil (TAS-102) (35 mg/m2/dose) was administered orally in continuous 28-day treatment cycles until a discontinuation criterion was met. One treatment cycle of TAS-102 (35mg/m2/dose) involved administration of dose twice per day, after morning and evening meals, for 5 days a week, with 2 rest days, for 2 weeks, followed by a 14-day rest period. Survival follow-up could be extended until the target number of events (288 deaths) was reached.
- Placebo: placebo was administered orally in continuous 28-day treatment cycles until a discontinuation criterion was met. One treatment cycle of placebo involved administration of dose twice per day, after morning and evening meals, for 5 days a week, with 2 rest days, for 2 weeks, followed by a 14-day rest period. Survival follow-up could be extended until the target number of events (288 deaths) was reached.
Period: Overall Study
Arm/Group | TAS-102（Trifluridine/Tipiracil） | Placebo
Started | 271 | 135
Completed | 271 | 135
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TAS-102（Trifluridine/Tipiracil）: TAS-102 (35 mg/m2/dose) was administered orally in continuous 28-day treatment cycles until a discontinuation criterion was met. One treatment cycle of TAS-102 (35mg/m2/dose) involved administration of dose twice per day, after morning and evening meals, for 5 days a week, with 2 rest days, for 2 weeks, followed by a 14-day rest period. Survival follow-up could be extended until the target number of events (288 deaths) was reached.
- Total: Total of all reporting groups
Arm/Group | TAS-102（Trifluridine/Tipiracil） | Placebo | Total
Number analyzed (Participants) | 271 | 135 | 406
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 206 | 103 | 309
  >=65 years | 65 | 32 | 97
Age, Continuous [Median (Full Range); unit: years] | 58 [26 to 81] | 56 [24 to 80] | 57 [24 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 51 | 152
  Male | 170 | 84 | 254
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 271 | 134 | 405
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 271 | 135 | 406
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 55 | 26 | 81
  China | 204 | 101 | 305
  Thailand | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival（OS）
Description: The primary endpoint was Overall Survival (OS), which was defined as the time from random assignment to the date of death. In the absence of confirmation of death or for patients alive at the OS cutoff date, survival time was censored at the date of last trial follow-up or the cutoff date, whichever was earlier.
Time Frame: Every 8 weeks. Survival status should be collected for up to 12 months after the last patient is randomized or until the target number of events (deaths) is met, whichever is later.
Population: The intent-to-treat (ITT) population: the ITT population was comprised of all patients who were randomized to study medication.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TAS-102（Trifluridine/Tipiracil） | Placebo
Number analyzed (Participants) | 271 | 135
Months | 7.8 [7.1 to 8.8] | 7.1 [5.9 to 8.2]
Statistical Analysis 1: Comparison: TAS-102（Trifluridine/Tipiracil） vs Placebo; Test type: Superiority; p = 0.035, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.62 to 0.99]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Tumor assessments were performed throughout the study period and analyzed using Response Evaluation Criteria in Solid Tumors criteria (Version 1.1, 2009). Progression-free survival was defined as the time (in months) from the date of randomization until the date of the Investigator-assessed radiological disease progression or death due to any cause. Patients who received non-study cancer treatment before radiologic evidence of disease progression were censored at the date of the last evaluable tumor assessment before initiation of non-study cancer treatment.
Time Frame: Every 8 weeks. Tumor assessments will be performed until radiologic progression develops or the start of new anticancer treatment, for up to 12 months after the last patient is randomized or until the target number of events (deaths) is met.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TAS-102（Trifluridine/Tipiracil） | Placebo
Number analyzed (Participants) | 271 | 135
Months | 2.0 [1.9 to 2.8] | 1.8 [1.7 to 1.8]
Statistical Analysis 1: Comparison: TAS-102（Trifluridine/Tipiracil） vs Placebo; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.43, 95% CI 2-sided [0.34 to 0.54]

3. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Time to treatment failure was defined as the time (in months) from the date of randomization until the date of radiologic disease progression, permanent discontinuation of study treatment, or death due to any cause. Censoring for TTF was also applied for those patients who were given non-study cancer treatment, with censoring at the time when the patient began the non-study cancer treatment.
Time Frame: From randomization until the date of radiologic disease progression, permanent discontinuation of study treatment, or death due to any cause, assessed up to 30 months.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS-102（Trifluridine/Tipiracil） | Placebo
Number analyzed (Participants) | 271 | 135
months | 1.9 [1.9 to 2.2] | 1.8 [1.7 to 1.8]
Statistical Analysis 1: Comparison: TAS-102（Trifluridine/Tipiracil） vs Placebo; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.37 to 0.58]

4. Secondary Outcome: Overall Response Rate (ORR; Complete Response [CR] or Partial Response [PR] Using RECIST Criteria)
Description: The assessment of ORR was based on Investigator review of the images according to RECIST Version 1.1. Overall response rate was defined as the proportion of patients with objective evidence of complete response (CR) or partial response (PR). At the analysis stage, the best overall response was assigned for each patient as the best response recorded from all responses recorded after study randomization. If applicable, responses recorded after disease progression or initiation of non-study cancer treatment was excluded. A patient's best response assignment of stable disease (SD) needed to be maintained for at least 6 weeks after study randomization. If a patient didn't meet this condition, best response was assigned "Not evaluable".
Time Frame: as for outcome 3
Population: The tumor response evaluable (TR) population: the TR population included all patients in the ITT population who had measurable disease (at least 1 target lesion) at baseline and with at least 1 tumor evaluation while on treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAS-102（Trifluridine/Tipiracil） | Placebo
Number analyzed (Participants) | 261 | 130
percentage of participants | 1.1 [0.2 to 3.3] | 0.0 [0.0 to 2.8]
Statistical Analysis 1: Comparison: TAS-102（Trifluridine/Tipiracil） vs Placebo; Test type: Superiority; p = 0.554, Fisher Exact; Difference in ORR = 1.1, 95% CI 2-sided [-0.1 to 2.4]

5. Secondary Outcome: Disease Control Rate (DCR; CR, PR, or Stable Disease)
Description: The assessment of DCR paralleled that of ORR, with DCR defined as the proportion of patients with objective evidence of CR, PR, or SD.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TAS-102（Trifluridine/Tipiracil） | Placebo
Number analyzed (Participants) | 261 | 130
percentage of participants | 44.1 [37.9 to 50.3] | 14.6 [9.0 to 21.9]
Statistical Analysis 1: Comparison: TAS-102（Trifluridine/Tipiracil） vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact; Difference in DCR = 29.4, 95% CI 2-sided [20.9 to 38.0]

6. Secondary Outcome: Duration of Response
Description: Duration of response was derived for those patients with objective evidence of PR or CR. Duration of response was defined as the time from the first documentation of response (CR or PR) to the first documentation of objective tumor progression or to death due to any cause. Patients alive and progression free as of the analysis cut-off date were censored at their last evaluable tumor response assessment prior to initiation of any non-study cancer treatment.
Time Frame: as for outcome 3
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TAS-102（Trifluridine/Tipiracil） | Placebo
Number analyzed (Participants) | 261 | 130
Months | 6.6 [3.9 to 9.2] | 0 [0 to 0]
Statistical Analysis 1: Comparison: TAS-102（Trifluridine/Tipiracil） vs Placebo; Test type: Superiority; p < 0.001, Fisher Exact; Odds Ratio (OR) = 29.4, 95% CI 2-sided [20.9 to 38.0]

7. Secondary Outcome: Safety and Tolerability Evaluation Will Focus on Adverse Events and Laboratory Assessments（Adverse Events）
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-related AEs were events between administration of study drug and up to 30 Days that were absent before treatment or that worsened relative to pre-treatment state. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability /incapacity; congenital anomaly. The AEs were graded for severity using National Cancer Institute Common Terminology Criteria for AEs.
Time Frame: From the time a patient signed informed until 30 day safety follow-up visit or until initiation of new anticancer treatment, or assessed up to 30 months.
Population: The as-treated (AT) population: the AT population contained all patients in the ITT population who received at least 1 dose of study medication and patients were analyzed according to treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-102（Trifluridine/Tipiracil） | Placebo
Number analyzed (Participants) | 271 | 135
Participants
  No AEs | 2 | 15
  One or more AEs | 269 | 120
  One or more TEAEs | 269 | 118
  TEAE severity by CTCAE grade:Grade1 | 23 | 32
  TEAE severity by CTCAE grade:Grade2 | 84 | 41
  TEAE severity by CTCAE grade:Grade3 | 127 | 33
  TEAE severity by CTCAE grade:Grade4 | 30 | 11
  TEAE severity by CTCAE grade:Grade5 | 5 | 1
  TEAE causality(Related) | 244 | 70
  TEAE causality(Not Related) | 25 | 48
  One or more TEAEs leading to discontinuation | 27 | 13
  One or more SAEs | 63 | 32
  One or more TESAEs | 63 | 31
  One or more TEAEs leading to death | 5 | 1

8. Secondary Outcome: Safety and Tolerability Evaluation Will Focus on Adverse Events and Laboratory Assessments（Laboratory Assessments）
Description: All laboratory values that were out of the normal range were to be evaluated for their clinical significance before exposing the patient to the next dose of study medication. Any laboratory abnormality that was clinically significant, e.g., results in delay of study medication dosing, study discontinuation, required treatment due to abnormal values, or was considered by the Investigator to be medical important, were to be reported as an AE, unless it was considered part of clinical manifestations to a clinical diagnosis that has already been reported as an AE.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | TAS-102（Trifluridine/Tipiracil） | Placebo
Number analyzed (Participants) | 271 | 135
Participants
  Anemia：Any Grade | 209 | 52
  Anemia：Grade >=3 | 48 | 8
  Leukopenia：Any Grade | 190 | 4
  Leukopenia：Grade >=3 | 56 | 0
  Neutropenia：Any Grade | 182 | 1
  Neutropenia：Grade >=3 | 90 | 0
  Lymphopenia：Any Grade | 146 | 34
  Lymphopenia：Grade >=3 | 39 | 3
  Thrombocytopenia：Any Grade | 96 | 10
  Thrombocytopenia：Grade >=3 | 8 | 2
  Lymphocytosis：Any Grade | 4 | 1
  Lymphocytosis：Grade >=3 | 1 | 0
  Increase in alkaline phosphatase level：Any Grade | 91 | 58
  Increase in alkaline phosphatase level：Grade >=3 | 11 | 5
  Hyperglycemia：Any Grade | 98 | 50
  Hyperglycemia：Grade >=3 | 7 | 3
  Increase in total bilirubin level：Any Grade | 99 | 28
  Increase in total bilirubin level：Grade >=3 | 19 | 10
  Hypoalbuminemia：Any Grade | 78 | 44
  Hypoalbuminemia：Grade >=3 | 8 | 0
  Hyponatremia：Any Grade | 81 | 38
  Hyponatremia：Grade >=3 | 12 | 6
  Hypocalcemia：Any Grade | 77 | 33
  Hypocalcemia：Grade >=3 | 3 | 1
  Increase in AST level：Any Grade | 63 | 40
  Increase in AST level：Grade >=3 | 10 | 7
  Increase in ALT level：Any Grade | 48 | 29
  Increase in ALT level：Grade >=3 | 3 | 4
  Hypokalemia：Any Grade | 31 | 11
  Hypokalemia：Grade >=3 | 2 | 1
  Increase in creatinine level：Any Grade | 13 | 10
  Increase in creatinine level：Grade >=3 | 3 | 0
  Hyperkalemia：Any Grade | 11 | 10
  Hyperkalemia：Grade >=3 | 1 | 0
  Hypercalcemia：Any Grade | 8 | 1
  Hypercalcemia：Grade >=3 | 0 | 1

9. Secondary Outcome: Overall Survival（OS）(Wild Type KRAS)
Description: The primary end point was OS, which was defined as the time from random assignment to the date of death. In the absence of confirmation of death or for patients alive at the OS cutoff date, survival time was censored at the date of last trial follow-up or the cutoff date, whichever was earlier.
  The OS indicated above as secondary outcome was analyzed by wild type KRAS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS-102（Trifluridine/Tipiracil） | Placebo
Number analyzed (Participants) | 271 | 135
months | 8.6 [7.4 to 10.9] | 7.4 [5.6 to 9.2]
Statistical Analysis 1: Comparison: TAS-102（Trifluridine/Tipiracil） vs Placebo; Test type: Superiority; p = 0.083, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.57 to 1.04]

10. Secondary Outcome: Overall Survival（OS）(Mutant Type KRAS)
Description: The primary end point was OS, which was defined as the time from random assignment to the date of death. In the absence of confirmation of death or for patients alive at the OS cutoff date, survival time was censored at the date of last trial follow-up or the cutoff date, whichever was earlier.
  The OS indicated above as secondary outcome was analyzed by mutant type KRAS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS-102（Trifluridine/Tipiracil） | Placebo
Number analyzed (Participants) | 271 | 135
months | 7.0 [5.4 to 8.0] | 6.5 [4.6 to 7.6]
Statistical Analysis 1: Comparison: TAS-102（Trifluridine/Tipiracil） vs Placebo; Test type: Superiority; p = 0.228, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.57 to 1.20]

11. Secondary Outcome: Progression-free Survival (PFS) (Wild Type KRAS)
Description: Progression-free survival was defined as the time (in months) from the date of randomization until the date of the Investigator-assessed radiological disease progression or death due to any cause. Patients who received non-study cancer treatment before radiologic evidence of disease progression were censored at the date of the last evaluable tumor assessment before initiation of non-study cancer treatment. The PFS indicated above as secondary outcome was analyzed by wild type KRAS.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | TAS-102（Trifluridine/Tipiracil） | Placebo
Number analyzed (Participants) | 271 | 135
months | 2.0 [1.9 to 3.4] | 1.8 [1.7 to 1.8]
Statistical Analysis 1: Comparison: TAS-102（Trifluridine/Tipiracil） vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.32 to 0.59]

12. Secondary Outcome: Progression-free Survival (PFS) (Mutant Type KRAS)
Description: Progression-free survival was defined as the time (in months) from the date of randomization until the date of the Investigator-assessed radiological disease progression or death due to any cause. Patients who received non-study cancer treatment before radiologic evidence of disease progression were censored at the date of the last evaluable tumor assessment before initiation of non-study cancer treatment. The PFS indicated above as secondary outcome was analyzed by mutant type KRAS.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | TAS-102（Trifluridine/Tipiracil） | Placebo
Number analyzed (Participants) | 271 | 135
Months | 2.2 [1.9 to 3.4] | 1.8 [1.7 to 1.9]
Statistical Analysis 1: Comparison: TAS-102（Trifluridine/Tipiracil） vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.31 to 0.65]

ADVERSE EVENTS:
Time Frame: Safety monitoring continued from the time a patient signed informed until 30 days after the last dose of study medication or until the initiation of another cancer therapy, whichever came first, up to 30 months.
Description: An AE was any untoward medical condition that occurred in a patient while participating in a clinical study and did not necessarily have a causal relationship with the use of the product. Treatment-emergent adverse events (TEAEs) were AEs that occurred from the initiation of any study medication administration and did not necessarily have a causal relationship to the use of the study medication.
Arm/Group | TAS-102 | Placebo
All-Cause Mortality (participants affected / at risk) | 205/271 | 111/135
Serious Adverse Events (participants affected / at risk) | 63/271 | 32/135
Other Adverse Events (participants affected / at risk) | 269/271 | 120/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS-102 (N=271) | Placebo (N=135)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Granulocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 3 (3)
Duodenal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 4 (4)
Intestinal obstruction (Gastrointestinal disorders) | 3 (4) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (7) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (4) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 2 (2) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 3 (3) | 0 (0)
Liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Azotaemia (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAS-102 (N=271) | Placebo (N=135)
Anaemia (Blood and lymphatic system disorders) | 124 (151) | 27 (28)
Neutropenia (Blood and lymphatic system disorders) | 98 (214) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 47 (94) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 23 (46) | 4 (5)
Nausea (Gastrointestinal disorders) | 104 (164) | 20 (25)
Vomiting (Gastrointestinal disorders) | 60 (96) | 13 (20)
Diarrhoea (Gastrointestinal disorders) | 54 (81) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 31 (40) | 24 (29)
Constipation (Gastrointestinal disorders) | 25 (33) | 20 (26)
Abdominal distension (Gastrointestinal disorders) | 23 (26) | 9 (9)
Dyspepsia (Gastrointestinal disorders) | 15 (19) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 10 (12) | 7 (9)
Fatigue (General disorders) | 69 (92) | 20 (20)
Asthenia (General disorders) | 29 (35) | 11 (11)
Pyrexia (General disorders) | 18 (20) | 10 (12)
Upper respiratory tract infection (Infections and infestations) | 14 (17) | 3 (5)
White blood cell count decreased (Investigations) | 102 (233) | 3 (3)
Neutrophil count decreased (Investigations) | 75 (191) | 0 (0)
Blood bilirubin increased (Investigations) | 53 (77) | 12 (13)
Aspartate aminotransferase increased (Investigations) | 33 (40) | 20 (20)
Platelet count decreased (Investigations) | 42 (75) | 2 (2)
Alanine aminotransferase increased (Investigations) | 25 (32) | 16 (17)
Blood alkaline phosphatase increased (Investigations) | 21 (22) | 15 (15)
Bilirubin conjugated increased (Investigations) | 17 (30) | 4 (4)
Haemoglobin decreased (Investigations) | 18 (20) | 3 (5)
Gamma-glutamyltransferase increased (Investigations) | 10 (10) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 81 (105) | 22 (25)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 14 (14) | 13 (13)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (16) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (7) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (18) | 13 (13)
Dizziness (Nervous system disorders) | 25 (34) | 6 (6)
Headache (Nervous system disorders) | 14 (15) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 10 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other